CLINICAL TRIAL: NCT06698783
Title: Practical Application and Evaluation of Fortimel Taste Optimization Nutritional Support in Oncology Patients: a Multicenter Real-World Study
Brief Title: Practical Application and Evaluation of Fortimel in Oncology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K6287
Record Dates: First submitted 2024-08-15; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Dietary Supplement: Fortimel

INTERVENTIONS:
Dietary Supplement: Fortimel — In this study, patients will be provided with ONS preparation (4 kinds of ready-to-drink special medical food) free of charge during the treatment period. Doctors will provide patients with different flavor nutritional preparations on a weekly basis, 2 bottles per day for patients with 1 flavor per week, and 14 bottles per day for each of 4 flavors at the recommended dosage of 400 kcal per day 28 days

SUMMARY:
This study is a multicenter registry and is a prospective, observational, real-world study.

Subjects were selected by clinicians for oral ONS nutritional intervention according to the actual clinical situation and the patient's wishes, and the observation period was 4 weeks.

Subjects will receive a ready-to-drink marketed formula for special medical purposes with 4 flavors for free Food liquid preparation (Nengli Yijia, Nutricia in the Netherlands) for rounds of nutritional intervention, providing

1 flavor per week, 1-2 bottles per day, 4 flavors for a total of 28 days. The basic nutritional status and quality of life of patients were mainly evaluated at multiple time nodes before and after nutritional intervention.

In order to improve the compliance of subjects, the all-round guardian platform (hereinafter referred to as the platform) by the China Initial Insurance Foundation was used during the intervention period to provide basic nutrition supervision, education and dietary guidance in routine nutrition support.

Recruitment method: Convenient sampling method is adopted, from the beginning of recruitment to the target sample size.

Follow-up period: After the start of the intervention, it will be carried out according to the plan of the follow-up task to the end of the intervention on the 28th day. The last telephone follow-up visit will complete on the 60th day after the end of the pre-end.

ELIGIBILITY:
Inclusion Criteria:

* Patients signed informed consent and volunteered to participate in the study
* Patients diagnosed with colorectal cancer or primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring, undifferentiated adenocarcinoma) or NSCLC stage I-iv. by histopathological examination of primary biopsy
* Cancer patients who were receiving chemoradiotherapy or immunotherapy were given 2 points for nutritional risk screening, and patients who met the conditions of ONS nutrition intervention were voluntarily enrolled to receive ONS nutrition intervention with Nertronecar
* Basic reading and communication skills
* The expected survival time is greater than 6 months

Exclusion Criteria:

* Combined cognitive dysfunction, mental disorder, impaired consciousness or unwillingness to partner
* Contraindications with chemotherapy or immunotherapy
* Prolonged bed rest, hemiplegia, or coma
* Intolerance of allergies to nutrients or their main components, such as lactose or galactose
* In the case of severe gastrointestinal symptoms of liver and kidney dysfunction, the serum creatinine glutamic pyruvic transaminase glutamic oxalacetic transaminase increases by more than 2.5 times, and the fasting blood glucose is over10mmol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
weight | One week before intervention and day 1, day 14 and day 28 of intervention.
  weight measured by body composition analyzer
fat-free mass index | One week before intervention and day 1, day 7,day 14,day 21, and day 28 of intervention.
  fat-free mass index measured by body composition analyzer
skeletal muscle index | One week before intervention and day 1, day 7, day 14, day 21, and day 28 of intervention.
  skeletal muscle index measured by body composition analyzer
food intake change | One week before intervention and day 1, day 7, day 14, day 21, and day 28 of intervention.
  calculated from recorded food intake through an online tool

SECONDARY OUTCOMES:
Satiety | Day 1, day 14,and day 28 of intervention
  VAS score
Gastrointestinal reactions | Day 1, day 14,and day 28 of intervention
  enteral nutrition tolerance scale tool
Adherence to nutritional formulations | Day 1, day 14,and day 28 of intervention
  using the patient's ONS compliance register
24h dietary intake | Day 1, day 14,and day 28 of intervention

OTHER OUTCOMES:
Major complications during treatment | 28 days since the intervention.
  General adverse reactions (dizziness, headache, fatigue and weakness, loss of appetite, nausea and vomiting, hair loss, dry mouth, dyspepsia, stomach discomfort, tissue edema, constipation, diarrhea, blood in the stool, etc.), nosocomial infection, respiratory failure, cardiovascular events (stroke, intracranial hemorrhage, cardiac arrest, myocardial infarction, etc.), radiation brain reactions, radiation pulmonary fibrosis, radiation pneumonitis, radiation pharyngitis, radiation esophagitis, radiation xerostomia, radiation otitis media, radiation mandibular arthritis, radiation neck skin atrophy, radiation caries, hearing loss, deafness, bone marrow suppression, endocrine disorders, pulmonary embolism, myocarditis, enteritis, acute pancreatitis, acute renal failure, gastrointestinal events (bleeding, intestinal perforation, acute pancreatitis, etc.) or a decrease of 10% or more from baseline by the Barthel index.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongcheng district，Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No